CLINICAL TRIAL: NCT00340782
Title: The Influence of Social and Environmental Factors on Fecundability in a Maya Community of Guatemala
Brief Title: Influence of Social and Environmental Factors on Women's Reproductive Function in a Maya Community of Guatemala
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999906145; 06-E-N145
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-04-21

CONDITIONS: Early Pregnancy
Keywords: Menstrual Cycles; Early Pregnancy; Reproductive Hormones; Stress; Adrenal Function

SUMMARY:
This study will explore the influence of social and environmental factors, such as stress, nutrition, health status, etc., on women's reproductive function.

Married Mayan women 16-42 years of age who live in the rural highlands of Guatemala and who have given birth to at least one child are eligible to participate in this study.

Participants are interviewed about their demographic, social, family, personal, health, reproductive and economic situations. They have saliva and urine samples collected three times a week for up to 1 year. Their nutritional and health status is assessed monthly.

DETAILED DESCRIPTION:
Background & Objectives: To explore the influence that social and environmental factors have on women's reproductive function. The general hypothesis is that deterioration in the quality of women's reproductive environment (e.g. psychosocial stress, nutritional status, health status, etc.) would have deleterious effects on fecundability and early pregnancy maintenance.

Study population: Data were collected from Mayan women in Guatemala. The reduced ethnic and socio-economic heterogeneity of this traditional population, as compared to that of an industrialized society, increased the robustness of the study design.

Inclusion and exclusion criteria: The goal was to evaluate fecundability and early pregnancy, thus, only women who met all six of the following criteria were recruited: (1) cohabitating with husband, (2), parity greater than or equal to 1 (to reduce the number of infertile participants), (3) being between 16-42 years of age (women aged greater than or equal to 16 are considered adults in this Mayan community. In fact, the first two pre-requisite to participate were that women were married and had given birth to at least one child), (4) not pregnant at the onset of the study (5) not using any form of contraception, and (6) last birth greater than six months prior to the onset of the study.

Human Subject Protection: Participants' recruitment was voluntary. Consent was obtained orally because most participants were illiterate, Privacy and confidentiality were assured, and participants were informed that they could discontinue their participation at any time with no cost or consequences to them. No deception, or covert observation, or interviewing of children were involved. I.D. numbers (not names) were used in recording the data. Names of participants are kept separately from data. All names and data files are kept in password protected NIEHS-computer or CDs stored under lock and key. Only ID numbers are used in analyses. Names are stored in case future research is needed. We have no current plants for research that involves re-contacting participants. Such research would entail a separate IRB application.

Design and outcome parameters: Saliva and first-morning urine specimens plus interview data were collected every other day, for a total of three times each week for up to one year. Participants' stress is measured via interview instruments as well as salivary and urinary free cortisol levels. Fecundability and early pregnancy are monitored through the determination of progesterone and estrone conjugates, luteinizing and follicle stimulating hormones, and chorionic gonadotropin. Nutritional and health assessments were achieved through standard medical and anthropometric procedures. Lactation, frequency and timing of intercourse, socio-economic status, and participant's life and reproductive history were all assessed via interview instruments. The data collection phase of this project is finished. Specimen and data analyses will continue including further assessment of stress, fecundability, and early pregnancy. Specimen analyses will be conducted by our collaborator Dr. Barry G. England at the University of Michigan under a separated University of Michigan IRB approval.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

Women who met all five of the following criteria were invited to participate: (1) cohabitating with husband, (2) not pregnant at the onset of the study, (3) parity greater than or equal to 1, (4) not using any form of contraception, and (5) last birth greater than six months prior to the onset of the study.

Ages: 16 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0
Dates: Start 2006-04-13; Study Completion 2008-04-21

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - NIEHS, Research Triangle Park, Research Triangle Park, North Carolina

REFERENCES:
- [Background] Neugebauer R, Kline J, Stein Z, Shrout P, Warburton D, Susser M. Association of stressful life events with chromosomally normal spontaneous abortion. Am J Epidemiol. 1996 Mar 15;143(6):588-96. doi: 10.1093/oxfordjournals.aje.a008789. PMID 8610676